CLINICAL TRIAL: NCT02339025
Title: The NCI-DoD TriCare Feasibility Study
Brief Title: DoD-NCI TRICARE Feasibility Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999915062; 15-C-N062
Record Dates: First submitted 2015-01-14; First posted 2015-01-15 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Cancer
Keywords: Cohort; Participation; Biobank
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Tricare Participants: From WRNMC

SUMMARY:
Background:

- Researchers at the National Cancer Institute and the Department of Defense are trying to learn more about what causes cancer, heart disease, and other health problems. To do this, they gather data on risk factors and biological markers. They get these data from large groups of people in long-running studies. As these groups of people age, researchers must form new groups. TRICARE is a health insurance program for uniformed service members and their families. It is a major part of the Military Health System. Researchers hope to form a new study group from TRICARE members. This study will test if TRICARE members will take part in a research study.

Objectives:

- To test if TRICARE members will take part in a research study.

Eligibility:

- TRICARE members aged 35 74 with military primary care providers at Walter Reed National Military Medical Center. They must not have a prior diagnosis of cancer other than non-melanoma skin cancer.

Design:

* Participants will fill out a survey. It will ask about their risk factors for cancer and other chronic diseases. Their medical records will be reviewed. They will give a blood sample.
* If a larger study is formed, then participants data will be used in the larger study. They may be asked to give more samples.

DETAILED DESCRIPTION:
DCEG has a long history of developing and running major cohort studies, and these form the

backbone of the research portfolio in the Division. Existing cohorts, including but not limited to

AARP, PLCO and USRT, have been extremely productive and have generated a wealth of

information about potential cancer risk factors and biological markers. In the next decade, these cohorts will reach the end of their natural lifetime due to the length of time since the baseline questionnaire, the average age of the participants, and the depletion of biological samples. There is the need, therefore, to start planning for the next generation of cohorts that will be able to continue to address current and future hypotheses about the etiology of cancer. A working group within DCEG was formed to discuss potential settings, and a cohort study within the US military setting was selected as one of the promising possibilities. Attractive features conducive to conducting a cohort study using the TriCare health insurance system was the possibility of linkage to numerous electronic databases, including those that maintain addresses and enrollment status, pharmacy databases, medical records databases, and cancer registry and mortality databases. Tricare is a health care insurance program for uniformed service members (active, Guard/Reserve, retired) and their families.

Our overarching, long-term, objective is to build a new prospective multi-center adult cohort

among the membership of the Tricare insurance plan. The cohort will have rich exposure

information and accurate outcome information that will be used as a Divisionwide resource to

investigate novel hypotheses about the etiology of cancer, using questionnaire data, medical

records, tumor tissue and serial biospecimens. Given the large-scale nature of the anticipated cohort study, we plan to begin the work by conducting a feasibility study at military treatment facility, Walter Reed National Medical Center (WRNMMC).

The goal of the feasibility study is to help us determine what will be possible in a larger effort.

Several other feasibility studies are being conducted by other groups in DCEG. Depending on the outcome of these studies, DCEG senior leadership will make a decision on whether one large cohort or several smaller cohorts should move forward.

The feasibility study will have two parts: Part 1) we will randomly select and invite to participate, by post, a stratified sample of 1,000 eligible beneficiaries aged 35-74 years old. All participants will be asked to access a study website, complete an on-line consent form which includes consent for access to electronic health records, complete an on-line questionnaire, and provide a blood specimen within three months of enrolling in the study. The letter will offer a paper-based option for consent and questionnaire completion for those unwilling or unable to access the website. The following outcomes will be evaluated: %

enrollment, % questionnaire completion, % agreement to blood draw, % completion of blood draws, the time between enrollment and blood draw, duration of enrollment in Tricare, % with

supplemental civilian insurance, feasibility of linking electronic patient databases to each other and to the questionnaire data, and available characteristics of the participants and the non-participants; Part 2) Using MDR files, the Defense Health Agency (DHA) will provide frequencies on place of cancer diagnosis and treatment (military treatment facility vs. civilian hospital) and availability of treatment data for eligible beneficiaries with a diagnosis of cancer other than nonmelanoma skin cancer within the past 12 months. No individual level data will be collected. The protocol is formatted for submission to the WRNMMC.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be selected according to the MTF, gender, age, and race/ethnicity. Beneficiaries aged 35-74 years with military primary care providers at WRNMMC or FBCH or beneficiaries living in these catchment or service areas.

EXCLUSION CRITERIA:

Beneficiaries less than 35 years of age will be excluded because cancer incidence at these ages is low and therefore it is unlikely to be feasible from a cost/information perspective to include them. Beneficiaries 75 years of age or older will be excluded because it is unlikely they will have long-term follow-up.

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants will be asked to access a study website, complete an on-line consent form which includes consent for access to electronic health records, complete an on-line questionnaire, and provide a blood specimen.
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2018-08-18 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Participation rates | End of study recruitment
  Participant rates
Data linkage | Before study recruitment
  Data linkage

SECONDARY OUTCOMES:
Cross-sectional biomarker study | End of study recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Schairer, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Walter Reed National Medical Center, Bethesda, Maryland, United States